CLINICAL TRIAL: NCT05952245
Title: The Effect of Instant Message-delivered Brief Cognitive Behavioural Therapy for Insomnia (CBT-I) in Stroke Family Caregivers: a Mixed Method Study
Brief Title: Instant Message-delivered Cognitive Behavioural Therapy for Insomnia (CBT-I)Stroke Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CBTI2023
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2023-06

CONDITIONS: Stroke; Insomnia; Depressive Symptoms; Caregiver Burnout; Psychological Distress; Mobile Phone Use
MeSH Terms: conditions — Stroke; Sleep Initiation and Maintenance Disorders; Depression; Caregiver Burden; Cell Phone Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Receiving CBT-I based EMI messages.
  Interventions: Behavioral: iCBTI-based EMI
- Control Group (Active Comparator): Receiving education-based EMI messages.
  Interventions: Behavioral: Education-based EMI

INTERVENTIONS:
Behavioral: iCBTI-based EMI — Including brief iCBT-I for sleep support, stroke care education, and nurse-led real-time chat-based support messages, which were delivered according to participants' preferences (e.g., time and frequency).
  Arms: Intervention Group
Behavioral: Education-based EMI — Stroke and brief sleep hygiene education with chat-based support on the topics.
  Arms: Control Group

SUMMARY:
The proposed trial aims to assess the effectiveness of Cognitive-behavioural therapy for insomnia (CBT-I) based ecological momentary intervention (EMI) for reducing insomnia symptoms among stroke caregivers.

DETAILED DESCRIPTION:
Existing studies reported that 40-95% of family caregivers had clinically significant insomnia symptoms including reduced total sleep duration, prolonged sleep onset latency, frequent night awakenings, and poor sleep efficiency and quality.

Cognitive-behavioural therapy for insomnia (CBT-I) has shown a large effect in reducing insomnia among adults. Innovative and interactive technologies, such as Internet-delivered CBT-I (iCBT-T), have therefore been incorporated into CBT-I, which was identified to have similar effects to that of traditional CBT-I.

In the proposed trial, screened stroke caregivers will be recruited from community centres, rehabilitation centres, and tertiary hospitals in HK. The intervention group will receive CBTI-based EMI through instant messaging applications as personalised and real-time psychological support led by nurses for 3 months. The control group will only receive stroke and brief sleep hygiene education with chat-based support on the topics.The primary outcomes are Sleep Condition Indicator (SCI) and Insomnia Severity Index (ISI) scores. Secondary outcomes will include sleep quality, depressive symptoms, anxiety symptoms, caregiver's burden, quality of life, and et al. A post-trial qualitative study will be conducted to understand the participants' experience of and compliance with the EMI.

ELIGIBILITY:
Inclusion Criteria:

* Primary family caregiver (Aged ≥18) of stroke survivor
* Able to read and communicate in Chinese
* Engaged caregiving roles for > 4 hours per day;
* Able to use a smartphone messaging app (e.g., WhatsApp and WeChat)
* SCI ≤ 21 scores (i.e., clinically significant insomnia)

Exclusion Criteria:

* Has provided care for <1 month prior to recruitment
* Has a diagnosis of psychiatric disease or is currently taking psychotropic drugs
* Currently taking medication to help with sleep
* Currently participating in any type of psychological intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Sleep Condition Indicator (SCI) | 24 weeks
  An eight-item rating scale that was developed to screen for insomnia disorder based on DSM-5 criteria. Possible total score ranges from 0 to 32, with higher values indicative of better sleep.
Insomnia Severity Index (ISI) | 24 weeks
  A 7-item scale with scoring ranging from 0-28, a higher score indicate more severe insomnia symptoms

SECONDARY OUTCOMES:
Sleep quality (Pittsburgh Sleep Quality Index [PSQI]) | 24 weeks
  A 19-item scale ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality
Depressive symptoms (Patient Health Questionnaire-9 [PHQ-9]): | 24 weeks
  A 9-item scale with score ranging from 0 to 27, higher scores indicate higher severity of depressive symptom
Anxiety symptoms (Generalized Anxiety Disorder-7 [GAD-7]) | 24 weeks
  A 7-item scale with score ranging from 0 to 21, higher scores indicate higher severity of anxiety symptom
Caregiver's burden (Zarit Burden Interview [ZBI-4]) | 24 weeks
  A 4-item scale with score ranging from 0 to 16, higher scores indicate higher severity of caregiving burden
Quality of life (EuroQol 5-dimension 5-level questionnaire [EQ-5D-5L]) | 24 weeks
  The EQ-5D-5L assesses five health dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each rated on five levels of severity, with scores ranging from -0.864 to 1, where higher scores indicate better quality of life.
  Additionally, it includes a visual analogue scale (VAS), ranging from 0 (the worst health imaginable) to 100 (the best health imaginable).
Positive experiences from caregiving (Positive Aspect of Caregiving [PAC]) | 24 weeks
  An 11-item scale with scores ranging from 0 to 44. A higher score indicates a more positive caregiving experience.
Caregiving self-efficacy (Caregiving Self-Efficacy Scale [CSES-8]) | 24 weeks
  An 8-item scale with scores ranging from 1 to 10, with higher scores indicating higher self-efficacy.
Sleep parameters (Consensus Sleep Diary Core Version) | 24 weeks
  The Consensus Sleep Diary Core Version will be used to collect sleep parameters (e.g., sleep efficiency and total sleep time).
Dysfunctional Beliefs and attitudes about Sleep (Dysfunctional Beliefs and attitudes about Sleep [DBAS]) | 24 weeks
  A 16-item scale with scores ranging from 0 to 160, with higher scores indicating greater dysfunctional beliefs about sleep.
Sleep hygiene statue (Sleep Hygiene Index [SHI]) | 24 weeks
  A 13-item scale with ratings from 0 to 52, where higher scores indicate poorer sleep hygiene status.
Sleep-related behavior (Chinese short-form of the sleep-related behavior questionnaire [SRBQ-SF]) | 24 weeks
  A 23-item scale with scores ranging from 0 to 92. A higher score indicates more sleep-related safety behaviors.
State of sleep effort (Glasgow Sleep Effort Scale [GSES]) | 24 weeks
  A 7-item scale with scores ranging from 0 to 14, where higher scores indicate greater effort to sleep over the past week.
Sleep-related quality of life (Glasgow Sleep Impact Index [GSII]) | 24 weeks
  The primary measureable outcomes for the GSII reflect VAS scores (0-100; with lower scores reflecting negative impact) for each of the three specified ranks, capturing impairment in the past two weeks.
  GSII reflect VAS scores (0-100; with lower scores reflecting negative impact) for each of the three
Feedback on iCBT-I intervention | 24 weeks
  Feedback on the sleep support programme will be collected, focusing on various aspects such as perceived usefulness and willingness to recommend the program. Each aspect will be evaluated using a 5-point Likert scale, where higher scores indicate more positive evaluations.
Adverse events | 24 weeks
  Feedback on adverse events related to the iCBT-I intervention, such as fatigue, will be collected.

CONTACTS AND LOCATIONS:
Locations (5):
- Hong Kong (5):
  - Hong Kong PHAB Association, Hong Kong
  - Hong Kong Stroke Association, Hong Kong
  - NT West Community Centre, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Hong Kong Society for Rehabilitation, Hong Kong